CLINICAL TRIAL: NCT04153565
Title: A Phase Ib Clinical Study to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) in Combination With Cisplatin and Pemetrexed in Treatment-naive Participants With Advanced Malignant Pleural Mesothelioma (KEYNOTE-A17).
Brief Title: A Study of Pembrolizumab in Combination With Cisplatin and Pemetrexed in Advanced Malignant Pleural Mesothelioma (MPM) (MK-3475-A17)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-A17; MK-3475-A17 (Other: Merck Protocol Number); 195054 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Mesothelioma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Mesothelioma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Cisplatin + Pemetrexed (Experimental): Pembrolizumab 200 mg IV every 3 weeks (Q3W) in combination with Cisplatin 75 mg/m^2 IV, and Pemetrexed 500 mg/m^2 IV for 4-6 cycles followed by monotherapy of Pembrolizumab up to 35 cycles from the first dose of the study in treatment phase (approximately 2 years).
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Participants will receive Pembrolizumab 200 mg IV every 3 weeks (Q3W) until disease progression, or until participant has received 35 administrations of Pembrolizumab (approximately 2 years).
  Other Names: Keytruda; MK-3475
Drug: Pemetrexed — Participants will receive Pemetrexed 500 mg/m^2 IV on Day 1 of each cycle up to 4-6 cycles where each cycle = 3 weeks
  Other Names: Alimta
Drug: Cisplatin — Participants will receive Cisplatin 75 mg/m^2 IV on Day 1 of each cycle up to 4-6 cycles where each cycle = 3 weeks
  Other Names: Platinol-AQ

SUMMARY:
This is a multicenter, open-label, non-randomized, study of pembrolizumab in combination with cisplatin and pemetrexed in treatment of naïve participants with a histologically confirmed diagnosis of advanced/unresectable malignant pleural mesothelioma (MPM) in Japanese participants. This study will evaluate the safety, tolerability, and preliminary efficacy of pembrolizumab in combination with cisplatin and pemetrexed. The primary objective is to evaluate the safety and tolerability of treatment with pembrolizumab in combination with cisplatin and pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of advanced/unresectable malignant pleural mesothelioma (MPM)
* Have at least one measurable disease, which is systemic therapy naïve, radiologically assessed by the local site investigator per modified Response Evaluation Criteria in Solid Tumors (RECIST) using imaging scanned within 28 days prior to the first dose in this study
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Has a life expectancy of at least 3 months
* Demonstrate adequate organ function
* Male participants are eligible to participate if they agree to remain abstinent or agree to use contraception unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, using contraceptives or is not a woman of child bearing potential (WOCBP)

Exclusion Criteria:

* A WOCBP who has a positive pregnancy test within 72 hours prior to treatment allocation
* Has received prior therapy with an anti-programmed cell-death 1 (anti PD-1), anti programmed cell-death ligand 1 (anti-PD-L1), or anti programmed cell-death ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has previously received systemic anti-cancer therapy (including investigational agents) for MPM
* Participants who received (neo) adjuvant previously may be eligible, only if the last dose of chemotherapy was completed at least 6 months before registration. Such participants must have recovered from all adverse events (AEs) due to previous (neo) adjuvant therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible
* Received radiation therapy to the lung that is > 30 gray (Gy) within 6 months of the first dose of trial treatment
* Completed palliative radiotherapy within 7 days of the first dose of trial treatment
* Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis
* Had a major surgery within 3 months prior to the first administration in this study
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction (≥Grade 3) to treatment a monoclonal antibody/components of the study intervention
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Is being treated for pericardial effusion, or has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions is eligible
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- Japan (4):
  - Hyogo College of Medicine Hospital ( Site 0003), Nishinomiya, Hyōgo
  - Kanagawa Cancer Center ( Site 0004), Yokohama, Kanagawa
  - JOHAS Okayama Rosai Hospital ( Site 0002), Okayama
  - National Cancer Center Hospital ( Site 0001), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kijima T, Kato T, Goto Y, Kuribayashi K, Mikami K, Negi Y, Murakami S, Yoshida T, Homma M, Wakana A, Noguchi K, Fujimoto N. KEYNOTE-A17: First-Line Pembrolizumab Plus Cisplatin-Pemetrexed in Japanese Participants With Advanced Pleural Mesothelioma. Cancer Sci. 2025 Aug;116(8):2208-2217. doi: 10.1111/cas.70082. Epub 2025 May 23. PMID 40407381
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Pemetrexed + Cisplatin: Participants received pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) in combination with pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV for 4-6 cycles, followed by pembrolizumab 200 mg/m^2 IV monotherapy Q3W for up to 35 cycles from the first dose of the study treatment (approximately 2 years). Each cycle was 21 days.
Period: Overall Study
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Started | 19
Completed | 6
Not Completed | 13
Not completed — Death | 13

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT) During Cycle 1, Per Common Terminology Criteria for Adverse Events (AEs), Version 5.0 (CTCAE)
Description: DLTs were assessed during Cycle 1 (21 days) and defined as any of the following, if considered by investigator to be related to any of the study interventions: Grade 4 hematologic toxicities, except neutropenia and febrile neutropenia; Grade 4 neutropenia lasting >7 days despite appropriate supportive treatment; Grade 4 febrile neutropenia only if the event considered as clinically significant by investigator and sponsor; any Grade 4 non-hematologic toxicity (except laboratory test abnormal including transient electrolyte abnormalities); any Grade 3 non-hematologic toxicity lasting >72 hours despite appropriate supportive treatment (not laboratory); and any Grade 4 laboratory test value abnormality; any Grade 3 laboratory test value abnormality lasting >7 days; delay in start of second course of more than 2 weeks (more than 35 days after the first dose) due to toxicity related to study procedures; any Grade 5 toxicity.
Time Frame: Up to 3 weeks (through Cycle 1 [21 days])
Population: All participants who received at least 1 dose of study intervention and who met the criteria for DLT evaluability by finishing Cycle 1 without a DLT or having experienced a DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 18
Participants | 2

2. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE.
Time Frame: Up to approximately 34 months
Population: All participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Participants | 19

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Participants | 6

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who have a Complete Response (CR: disappearance of target and non-target lesions and normalization of tumor markers) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions). ORR was based on modified Response Evaluation Criteria In Solid Tumors (RECIST) for Malignant Pleural Mesothelioma (MPM) as assessed by investigator.
Time Frame: Up to approximately 31 months
Population: All participants who received at least 1 dose of study intervention
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Percentage of participants | 73.7 [48.8 to 90.9]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had a Complete Response (CR: disappearance of target and non-target lesions and normalization of tumor markers) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.]) DCR was based on modified RECIST for MPM as assessed by investigator.
Time Frame: Up to approximately 31 months
Population: All participants who received at least 1 dose of study intervention
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Percentage of participants | 94.7 [74.0 to 99.9]

6. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrate a confirmed complete response (CR: disappearance of target and non-target lesions and normalization of tumor markers) or confirmed Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. DOR was based on modified RECIST for MPM as assessed by investigator.
Time Frame: Up to approximately 31 months
Population: All participants who received at least 1 dose of study intervention and demonstrated a confirmed response (CR or PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 14
Months | 16.8 [3.0 to NA] — NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse

ADVERSE EVENTS:
Time Frame: Up to approximately 34 months
Description: All-cause mortality table includes all allocated participants. Serious and other AEs include all participants who received at least 1 dose of study intervention. Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Pembrolizumab + Pemetrexed + Cisplatin
All-Cause Mortality (participants affected / at risk) | 13/19
Serious Adverse Events (participants affected / at risk) | 7/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Cisplatin (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Cisplatin (N=19)
Anaemia (Blood and lymphatic system disorders) | 11 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (13)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (15)
Diarrhoea (Gastrointestinal disorders) | 10 (12)
Lip dry (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (21)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Malaise (General disorders) | 9 (11)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (10)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 7 (12)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (10)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Renal impairment (Renal and urinary disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (9)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vascular pain (Vascular disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04153565/Prot_SAP_000.pdf